CLINICAL TRIAL: NCT02224846
Title: Postmarketing Surveillance Study: A Randomized, Open-Label, 3-Month Interventional Study of Tadalafil Effectiveness (2.5 mg and 5 mg) and Long-Term Safety Administered Once Daily in Chinese Men With Erectile Dysfunction
Brief Title: A Study of Tadalafil (LY450190) in Chinese Men With Erectile Dysfunction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15382; H6D-GH-B022 (Other: Eli Lilly and Company)
Record Dates: First submitted 2014-08-20; First posted 2014-08-25 (Estimated); Results first posted 2017-10-27 (Actual); Last update posted 2019-09-23 (Actual); Status verified 2019-09

CONDITIONS: Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction | interventions — Tadalafil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2.5 mg/5 mg tadalafil (Experimental): 2.5 mg tadalafil orally once daily for 3 months (Period 1) and then 5 mg tadalafil orally once daily for 21 months (Period 2).
  Interventions: Drug: Tadalafil
- 5 mg tadalafil (Experimental): 5 mg tadalafil orally once daily for 24 months (Period 1 and Period 2).
  Interventions: Drug: Tadalafil

INTERVENTIONS:
Drug: Tadalafil — Administered orally
  Other Names: LY450190

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of the study drug, taken once daily, known as tadalafil in Chinese participants with erectile dysfunction (ED). The study will last about up to 25 months for each participant.

ELIGIBILITY:
Inclusion Criteria:

* Have a history of erectile dysfunction for at least 3 months.
* Are sexually active and willing to remain sexually active with the same female partner during the study.
* Are willing to have 4 or more attempts of sexual intercourse with female partner between screening and first treatment start day.
* Are willing to stay away from any other medicines that the participants were already taking for erectile dysfunction during this study period.

Exclusion Criteria:

* Have erectile dysfunction, which is caused by any other primary sexual disorder.
* Have certain problems with kidneys, liver, heart, blood sugar levels, eyes, or central nervous system (study doctor will discuss with participants).
* Have a penis deformity or penile implant that in the opinion of the participants' doctor is significant.
* Have human immunodeficiency virus (HIV) infection.
* Are using certain kinds of medicines, which are not allowed in this study.
* Are allergic to tadalafil.
* Are planning to father a baby or are in a relationship with a pregnant partner.
* Are participating or discontinued participation in the past 30 days from any another clinical trial, which is not compatible with this trial.
* Have participated or discontinued from any other tadalafil clinical trial.
* Have a history of drug, alcohol, or substance abuse within the past 6 months.

Ages: 22 Years to 69 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 635 (Actual)
Dates: Start 2014-10; Primary Completion 2016-05 (Actual); Study Completion 2017-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (16):
- China (16):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Beijing
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Changchun
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Changsha
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chengdu
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chongqing
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fuzhou
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Guangzhou
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hangzhou
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hefei
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nanjing
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Qingdao
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Shanghai
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Suzhou
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wenzhou
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wuhan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Yinchuan

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement
URL: https://vivli.org/

RESULTS

PARTICIPANT FLOW:
Period: Period 1 (Month 3)
Arm/Group | 2.5 mg/5 mg Tadalafil | 5 mg Tadalafil
Started | 211 | 424
Received at Least One Dose of Study Drug | 210 | 421
Completed | 192 | 388
Not Completed | 19 | 36
Not completed — Adverse Event | 2 | 1
Not completed — Lost to Follow-up | 3 | 8
Not completed — Protocol Violation | 4 | 8
Not completed — Withdrawal by Subject | 8 | 18
Not completed — Sponsor Decision | 2 | 1
Period: Period 2 (Month 3 to Month 12)
Arm/Group | 2.5 mg/5 mg Tadalafil | 5 mg Tadalafil
Started | 192 | 388
Completed | 173 | 357
Not Completed | 19 | 31
Not completed — Adverse Event | 1 | 2
Not completed — Lost to Follow-up | 3 | 5
Not completed — Protocol Violation | 0 | 3
Not completed — Withdrawal by Subject | 15 | 19
Not completed — Physician Decision | 0 | 2
Period: Period 2 (Month 12 to Month 24)
Arm/Group | 2.5 mg/5 mg Tadalafil | 5 mg Tadalafil
Started | 173 | 357
Completed | 131 | 283
Not Completed | 42 | 74
Not completed — Adverse Event | 3 | 4
Not completed — Death | 1 | 0
Not completed — Lost to Follow-up | 7 | 13
Not completed — Protocol Violation | 4 | 11
Not completed — Withdrawal by Subject | 25 | 43
Not completed — Physician Decision | 0 | 2
Not completed — Sponsor Decision | 2 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | 2.5 mg/5 mg Tadalafil | 5 mg Tadalafil | Total
Number analyzed (Participants) | 211 | 424 | 635
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.6 (11.11) | 44.1 (10.90) | 43.6 (10.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 211 | 424 | 635
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 211 | 424 | 635
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  China | 211 | 424 | 635

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Experiencing at Least One Treatment Emergent Adverse Event (Serious or Non-Serious)
Description: A Treatment Emergent Adverse Event (TEAE) was defined as an event that first occurs or worsens (increases in severity) after baseline, regardless of causality or severity. The percentage of participants with TEAEs was calculated by dividing the number of participants with at least 1 TEAE over the 12-Month treatment period by the total number of participants analyzed, multiplied by 100%. A summary of serious and other non-serious adverse events, regardless of causality, is located in the Reported Adverse Events module.
Time Frame: Baseline through Month 12
Population: All enrolled participants who fulfill the study entry criteria and who receive at least one dose of tadalafil.
Measure: Number; unit: Percentage of participants
Arm/Group | 2.5 mg/5 mg Tadalafil | 5 mg Tadalafil
Number analyzed (Participants) | 210 | 421
Percentage of participants | 33.8 | 35.9

2. Primary Outcome: Percentage of Participants Experiencing at Least One Adverse Event Leading to Discontinuation
Description: Data presented are the number of participants who experienced 1 or more AEs (all causalities and drug-related) and serious AEs (SAEs) that lead to discontinuation. A summary of serious and other non-serious adverse events, regardless of causality, is located in the Reported Adverse Events module.
Time Frame: Baseline through Month 12
Population: All enrolled participants who fulfill the study entry criteria and who receive at least one dose of tadalafil.
Measure: Number; unit: percentage of participants
Arm/Group | 2.5 mg/5 mg Tadalafil | 5 mg Tadalafil
Number analyzed (Participants) | 210 | 421
percentage of participants | 1.4 | 0.7

3. Secondary Outcome: Change From Baseline in the International Index of Erectile Function- Erectile Function (IIEF-EF) Domain Questionnaire Score
Description: IIEF- EF is the sum of Questions 1-5 and 15 of the IIEF. Questions 1-5 are scored 0 (no sexual activity for Question 1, no sexual stimulation for Question 2 and did not attempt intercourse for Questions 3-5) to 5 (high erectile function) and Question 15 is scored 1 (very low confidence) to 5 (very high confidence), for a total score ranging from 1 to 30. Higher scores represent better erectile function. Least Squares (LS) mean of the change from baseline is from Mixed effect Model Repeat Measurement (MMRM) model. The model included covariates baseline + visit + pooled investigator + baseline*visit, where participant is a random effect.
Time Frame: Baseline, Month 1; Baseline, Month 3
Population: All enrolled participants who fulfill the study entry criteria, receive at least one dose of tadalafil, and have both baseline and postbaseline data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 2.5 mg/5 mg Tadalafil | 5 mg Tadalafil
Number analyzed (Participants) | 203 | 414
units on a scale
  Month 1 | 4.5 (0.42) | 6.2 (0.28)
  Month 3: number analyzed (Participants) | 193 | 391
  Month 3 | 6.1 (0.44) | 7.4 (0.28)

4. Secondary Outcome: Change From Baseline in the IIEF-EF Domain Questionnaire Score of 5 mg Tadalafil Treatments
Description: as for outcome 3
Time Frame: Baseline, Month 6; Baseline, Month 12;Baseline, Month 18; Baseline, Month 24
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 2.5 mg/5 mg Tadalafil | 5 mg Tadalafil
Number analyzed (Participants) | 203 | 414
units on a scale
  Month 6: number analyzed (Participants) | 186 | 376
  Month 6 | 8.2 (0.38) | 7.9 (0.27)
  Month 12: number analyzed (Participants) | 177 | 361
  Month 12 | 8.1 (0.43) | 7.9 (0.27)
  Month 18: number analyzed (Participants) | 166 | 341
  Month 18 | 8.6 (0.39) | 8.3 (0.27)
  Month 24: number analyzed (Participants) | 156 | 326
  Month 24 | 8.6 (0.44) | 8.5 (0.28)

5. Secondary Outcome: Percentage of Participants With "Yes" Responses to Sexual Encounter Profile (SEP) Diary
Description: Participant-assessed diary has 5 questions(QI-Q5): 4 of the 5 questions were analyzed. Q2: successful penetration, Q3: successful intercourse, Q4: satisfied with erection, and Q5: satisfied with sexual experience) for each sexual encounter made over a specified period of time. SEP Q1-Q5 scores were determined as the percentage of 'Yes' responses to each of the 5 questions out of all sexual attempts recorded during the time period.
Time Frame: Month 1, Month 3
Population: All enrolled subjects who fulfill the study entry criteria, receive at least one dose of tadalafil, and have both baseline and postbaseline data.
Measure: Mean (Standard Deviation); unit: Percentage of participants
Arm/Group | 2.5 mg/5 mg Tadalafil | 5 mg Tadalafil
Number analyzed (Participants) | 203 | 412
Percentage of participants
  Q2: successful penetration,Month 1 | 81.3 (34.58) | 86.7 (27.58)
  Q2: successful penetration,Month 3: number analyzed (Participants) | 193 | 391
  Q2: successful penetration,Month 3 | 88.2 (28.55) | 91.7 (23.11)
  Q3: successful intercourse,Month 1 | 41.2 (41.48) | 49.5 (42.85)
  Q3: successful intercourse,Month 3: number analyzed (Participants) | 193 | 391
  Q3: successful intercourse,Month 3 | 55.7 (43.19) | 60.1 (42.39)
  Q4: satisfied with erection, Month 1 | 24.8 (35.62) | 35.5 (41.63)
  Q4: satisfied with erection, Month 3: number analyzed (Participants) | 193 | 391
  Q4: satisfied with erection, Month 3 | 39.9 (43.73) | 43.5 (43.46)
  Q5: satisfied with sexual experience,Month 1 | 20.4 (32.81) | 31.1 (40.50)
  Q5: satisfied with sexual experience,Month 3: number analyzed (Participants) | 193 | 391
  Q5: satisfied with sexual experience,Month 3 | 35.7 (41.93) | 39.2 (43.06)

6. Secondary Outcome: Percentage of Participants Achieving Normal Erectile Functioning
Description: Participants achieving a normal erectile functioning (defined as having an IIEF-EF Domain score of >=26) at Month 1 and Month 3.
Time Frame: Month 1, Month 3
Population: as for outcome 5
Measure: Number; unit: Percentage of partcipants
Arm/Group | 2.5 mg/5 mg Tadalafil | 5 mg Tadalafil
Number analyzed (Participants) | 210 | 421
Percentage of partcipants
  Month 1: number analyzed (Participants) | 203 | 414
  Month 1 | 22.2 | 30.9
  Month 3: number analyzed (Participants) | 193 | 391
  Month 3 | 31.6 | 37.6

7. Secondary Outcome: Percentage of Participants Achieving Normal Erectile Functioning of 5 mg Tadalafil Treatments
Description: Participants achieving a normal erectile functioning (defined as having an IIEF-EF Domain score of >=26) at Month 6 and Month 12.
Time Frame: Month 6, Month 12, Month 18, Month 24
Population: as for outcome 5
Measure: Number; unit: Percentage of participants
Arm/Group | 2.5 mg/5 mg Tadalafil | 5 mg Tadalafil
Number analyzed (Participants) | 210 | 421
Percentage of participants
  Month 6: number analyzed (Participants) | 186 | 376
  Month 6 | 38.2 | 42.3
  Month 12: number analyzed (Participants) | 177 | 361
  Month 12 | 44.1 | 43.5
  Month 18: number analyzed (Participants) | 166 | 341
  Month 18 | 44.6 | 43.7
  Month 24: number analyzed (Participants) | 156 | 326
  Month 24 | 45.5 | 48.2

8. Secondary Outcome: Percentage of Participants With "Yes" Responses to Global Assessment Questions (GAQ)1 and GAQ2
Description: Participants with "yes" responses to GAQ Question 1 (GAQ1) and GAQ Question 2 (GAQ2) of the GAQ questionnaire at Month 3 and Month 12.
  GAQ1: Has the treatment you have been taking during this study improved your erections? GAQ2: If yes, has the treatment improved your ability to engage in sexual activity?
Time Frame: Month 3, Month12, Month 24
Population: All randomized participants who had evaluable data for Global Assessment Questions (GAQ)1 and GAQ2.
Measure: Number; unit: percentage of participants
Arm/Group | 2.5 mg/5 mg Tadalafil | 5 mg Tadalafil
Number analyzed (Participants) | 211 | 424
percentage of participants
  Month 3: GAQ1: number analyzed (Participants) | 193 | 392
  Month 3: GAQ1 | 89.6 | 95.7
  Month 12: GAQ1: number analyzed (Participants) | 177 | 361
  Month 12: GAQ1 | 96.6 | 97.5
  Month 24: GAQ1: number analyzed (Participants) | 156 | 326
  Month 24: GAQ1 | 96.8 | 95.7
  Month 3: GAQ2: number analyzed (Participants) | 193 | 392
  Month 3: GAQ2 | 86.5 | 92.1
  Month 12: GAQ2: number analyzed (Participants) | 177 | 361
  Month 12: GAQ2 | 95.5 | 96.1
  Month 24: GAQ2: number analyzed (Participants) | 156 | 326
  Month 24: GAQ2 | 96.2 | 94.5

ADVERSE EVENTS:
Description: All the participants who received at least one dose of study drug.
Arm/Group | 2.5 mg/5 mg Tadalafil | 5 mg Tadalafil
Serious Adverse Events (participants affected / at risk) | 15/210 | 17/421
Other Adverse Events (participants affected / at risk) | 86/210 | 178/421
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2.5 mg/5 mg Tadalafil (N=210) | 5 mg Tadalafil (N=421)
Angina unstable (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Maculopathy (Eye disorders) | 1 (1) | 0 (0)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 2 (2) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic cyst (Hepatobiliary disorders) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Urethral stricture postoperative (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Ankylosing spondylitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal cyst (Renal and urinary disorders) | 1 (1) | 1 (1)
Ureterolithiasis (Renal and urinary disorders) | 1 (2) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Varicocele (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2.5 mg/5 mg Tadalafil (N=210) | 5 mg Tadalafil (N=421)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Angina unstable (Cardiac disorders) | 0 (0) | 1 (1)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1)
Hypertensive heart disease (Cardiac disorders) | 0 (0) | 1 (1)
Microvascular coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Atrial septal defect (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Cerumen impaction (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Eustachian tube dysfunction (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Excessive cerumen production (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Mixed deafness (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Thyroid mass (Endocrine disorders) | 0 (0) | 2 (2)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 1 (1)
Conjunctivitis allergic (Eye disorders) | 0 (0) | 1 (1)
Diabetic retinopathy (Eye disorders) | 0 (0) | 1 (1)
Dry eye (Eye disorders) | 1 (1) | 0 (0)
Eye disorder (Eye disorders) | 0 (0) | 1 (1)
Eye swelling (Eye disorders) | 1 (1) | 0 (0)
Ocular discomfort (Eye disorders) | 0 (0) | 1 (1)
Uveitis (Eye disorders) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 1 (1) | 2 (2)
Xerophthalmia (Eye disorders) | 0 (0) | 1 (2)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 3 (3)
Abdominal distension (Gastrointestinal disorders) | 2 (2) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 4 (6) | 4 (4)
Chronic gastritis (Gastrointestinal disorders) | 4 (4) | 3 (3)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dental caries (Gastrointestinal disorders) | 3 (4) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 5 (6)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 2 (2)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 3 (3)
Enteritis (Gastrointestinal disorders) | 2 (2) | 2 (2)
Gastric dilatation (Gastrointestinal disorders) | 1 (1) | 2 (2)
Gastric polyps (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 2 (2)
Gastritis (Gastrointestinal disorders) | 3 (3) | 8 (10)
Gastritis erosive (Gastrointestinal disorders) | 0 (0) | 3 (3)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 4 (5)
Gingival bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gingival swelling (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 3 (3)
Large intestine polyp (Gastrointestinal disorders) | 1 (1) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 1 (1) | 4 (4)
Nausea (Gastrointestinal disorders) | 0 (0) | 3 (3)
Tooth disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1) | 6 (6)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 3 (3) | 4 (4)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (2)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis chronic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Fatty liver alcoholic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Gallbladder polyp (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic cyst (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic steatosis (Hepatobiliary disorders) | 1 (1) | 2 (2)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Anal abscess (Infections and infestations) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 5 (6)
Chronic sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 1 (1) | 3 (3)
Conjunctivitis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Dermatophytosis (Infections and infestations) | 0 (0) | 1 (1)
Ear infection (Infections and infestations) | 0 (0) | 1 (1)
Epididymitis (Infections and infestations) | 0 (0) | 1 (1)
Folliculitis (Infections and infestations) | 0 (0) | 3 (3)
Gastroenteritis (Infections and infestations) | 1 (1) | 3 (3)
Gingivitis (Infections and infestations) | 1 (1) | 0 (0)
Helicobacter infection (Infections and infestations) | 1 (1) | 0 (0)
Hepatitis b (Infections and infestations) | 0 (0) | 1 (1)
Hordeolum (Infections and infestations) | 1 (1) | 0 (0)
Infected dermal cyst (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 2 (2) | 3 (4)
Laryngitis (Infections and infestations) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 1 (1)
Mumps (Infections and infestations) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 1 (1) | 4 (4)
Otitis media chronic (Infections and infestations) | 0 (0) | 1 (2)
Periodontitis (Infections and infestations) | 6 (6) | 3 (3)
Pharyngitis (Infections and infestations) | 3 (3) | 8 (8)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Pulpitis dental (Infections and infestations) | 1 (1) | 2 (2)
Respiratory tract infection (Infections and infestations) | 1 (1) | 3 (3)
Rhinitis (Infections and infestations) | 3 (3) | 5 (6)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Tinea cruris (Infections and infestations) | 0 (0) | 1 (1)
Tinea infection (Infections and infestations) | 0 (0) | 1 (1)
Tinea manuum (Infections and infestations) | 0 (0) | 1 (2)
Tinea pedis (Infections and infestations) | 0 (0) | 3 (3)
Tonsillitis (Infections and infestations) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 5 (5) | 21 (25)
Urinary tract infection (Infections and infestations) | 3 (3) | 2 (2)
Viral upper respiratory tract infection (Infections and infestations) | 18 (24) | 39 (48)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)
Electrical burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Foreign body (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Heat stroke (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Lip injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Peripheral nerve injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Alanine aminotransferase increased (Investigations) | 5 (5) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Blood cholesterol increased (Investigations) | 1 (1) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0)
Blood glucose increased (Investigations) | 1 (1) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 3 (3)
Blood pressure systolic increased (Investigations) | 0 (0) | 1 (1)
Blood triglycerides increased (Investigations) | 1 (1) | 2 (2)
Blood urea increased (Investigations) | 1 (1) | 1 (1)
Blood uric acid increased (Investigations) | 4 (4) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 2 (2) | 1 (1)
High density lipoprotein increased (Investigations) | 1 (1) | 0 (0)
Lipids increased (Investigations) | 1 (1) | 1 (1)
Low density lipoprotein increased (Investigations) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 1 (1)
White blood cell count increased (Investigations) | 0 (0) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Folate deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Gout (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 (1) | 4 (5)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (5)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Exostosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (5)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Vertebral lesion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (5)
Carotid arteriosclerosis (Nervous system disorders) | 1 (1) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral artery stenosis (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1)
Diabetic neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 3 (3) | 9 (9)
Head discomfort (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 13 (14)
Migraine (Nervous system disorders) | 0 (0) | 1 (1)
Poor quality sleep (Nervous system disorders) | 0 (0) | 1 (1)
Radiculopathy (Nervous system disorders) | 0 (0) | 1 (1)
Tension headache (Nervous system disorders) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 2 (2)
Vertebrobasilar insufficiency (Nervous system disorders) | 0 (0) | 1 (1)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 4 (4) | 1 (1)
Irritability (Psychiatric disorders) | 1 (1) | 0 (0)
Premature ejaculation (Psychiatric disorders) | 0 (0) | 1 (1)
Sleep disorder (Psychiatric disorders) | 2 (2) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 1 (1) | 0 (0)
Glomerulonephritis chronic (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 2 (4) | 1 (1)
Renal cyst (Renal and urinary disorders) | 2 (2) | 2 (2)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal mass (Renal and urinary disorders) | 0 (0) | 1 (1)
Urethral pain (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Balanoposthitis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 3 (3)
Epididymal cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Prostatitis (Reproductive system and breast disorders) | 7 (7) | 4 (4)
Testicular pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 5 (5)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Reflux laryngitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Eczema (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Papule (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Skin disorder (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Breast feeding (Social circumstances) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 1 (1) | 2 (2)
Hypertension (Vascular disorders) | 3 (3) | 8 (9)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days